CLINICAL TRIAL: NCT05110859
Title: PHENOMENOLOGICAL QUALITATIVE SURVEY ABOUT NURSES FIRST WORK EXPERIENCE DURING COVID-19 PANDEMIC AT PIACENZA HOSPITAL, ITALY
Brief Title: QUALITATIVE SURVEY ABOUT NURSES FIRST WORK EXPERIENCE DURING COVID-19 PANDEMIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Unita Sanitaria Locale di Piacenza (Other)
Responsible Party: Principal Investigator, Maurizio Beretta, RN, Azienda Unita Sanitaria Locale di Piacenza
Other Study IDs: Qual_NeoCOVID
Record Dates: First submitted 2021-11-05; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Quality of Life
Keywords: covid 19; first work experience; nurse
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (1):
- first work experience nurses
  Interventions: Other: in-depth individual interviews

INTERVENTIONS:
Other: in-depth individual interviews — in-depth individual interviews to explore their perspectives on their first work experience during covid-19 pandemic

SUMMARY:
During covid-19 pandemic an huge reorganization of all PiacenzaHospital was done to manage the increasing requests for hosptitalization.

New nurses had to face first work experience in full pandemic Emergency. Altough even before the pandemic, being a newly graduated nurses was described as a stressful and isolating experience , we can't find studies in the literatureconcerning newly graduated and newly hired nurses during the pandemic pediod.

The study purpose is to describe and analyze, trough a phenomenological research, the experience of these nurses.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* first work experience nurses after gratuation
* not opposed to partecipate to this study

Exclusion Criteria:

* refusing to partecipate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nurses
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
nurses satisfaction | 6 months
  to detect emotional impact

CONTACTS AND LOCATIONS:
Locations (1):
- Piacenza Nursing School, University of Parma,, Piacenza, PC, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Casella G, Beretta M, Costa F, Opizzi D, Pompini P, Posla S, Sanfratello R, Guasconi M, Merlini C. Experiences of newly hired nurses during the Covid-19 emergency: descriptive qualitative research. Acta Biomed. 2023 Jun 14;94(3):e2023168. doi: 10.23750/abm.v94i3.14343. PMID 37326265